CLINICAL TRIAL: NCT05791266
Title: Safety of Sticker Pad Containing Essential Oil Containing Lavender and Ylang-ylang Oil Attached to the Collar for Decrease Blood Pressure in Healthy Volunteer
Brief Title: Safety of Sticker Pad Containing Essential Oil Containing Lavender and Ylang-ylang Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC 22028-20
Record Dates: First submitted 2023-03-14; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sticker pads containing lavender and ylang ylang oil (Experimental): Sticker pads , size 160 mm2, were produced by a certified ISO 9001 manufacturer and contained 0.3% lavender oil and 0.7% ylang ylang oil. The sticker pad was attached to the shirts of healthy volunteers for 2 hours. The outcomes were evaluated before, during and 30 minutes after removal of the pad.
  Interventions: Device: Sticker pads containing lavender and ylang ylang oil

INTERVENTIONS:
Device: Sticker pads containing lavender and ylang ylang oil — Sticker pads , size 160 mm2, were produced by a certified ISO 9001 manufacturer and contained 0.3% lavender oil and 0.7% ylang ylang oil. The sticker pad was attached to the shirts of healthy volunteers for 2 hours. The outcomes were evaluated before, during and 30 minutes after removal of the pad.

SUMMARY:
The aims of the study were to evaluate safety of sticker pads containing lavender and ylang ylang oil in healthy volunteers.

DETAILED DESCRIPTION:
The lavender and ylang ylang oil pad was attached to the shirts of healthy volunteers for 2 hours. The outcomes were evaluated before, during and 30 minutes after removal of the pad. Adverse reactions, irritation score, and quality of life were assessed. Blood pressure and pulse rate were also measured

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 60 years
* no allergic history of lavender and ylang ylang oil
* no dermatological diseases, immunocompromised diseases, seizures, asthma, or respiratory diseases.

Exclusion Criteria:

* an unstable condition of other diseases
* olfactory problems
* pregnancy
* lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Adverse reactions of the respiratory tract, skin, eye, and central nervous system | 2 hours
  The severity scores were 0 (no symptoms) to 3 (severe symptoms)

SECONDARY OUTCOMES:
Irritation of eye, respiratory, other neurological, and toxicity reaction | 2 hours
  Using a 0 to 100 scale, following an increase of severity
Systolic blood pressure | 2 hours
  Measure systemic blood pressure in mmHg
Diastolic blood pressure | 2 hours
  Measure diastolic blood pressure in mmHg
Pulse rate | 2 hours
  Measure pulse rate in beats/minutes
Rhinoconjunctivitis quality of life questionnaire | 2 hours
  Using a score of 1 (no problems) to 5 (severe problem)

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Study Director — Chulalongkorn University
Locations (1):
- Chulalongkorn Hospital, Bangkok, Thailand